CLINICAL TRIAL: NCT05480371
Title: Role of Cough Assist Device in Mechanically Ventilated Patients in Respiratory Intensive Care Unit : Assiut University Experience
Brief Title: Cough Assist Device in Mechanically Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hadeer Sayed Khalifa, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: cough assist device
Record Dates: First submitted 2022-07-18; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Mechanically Ventilated Patients

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional endotracheal suctioning (Active Comparator): Tracheal suctioning will be performed following the American Association for Respiratory Care recommendations: closed suction system, suction catheter with maximal internal-to-external diameter ratio of 0.5, delivery of 100% oxygen 30 s immediately before and 1 min after the procedure, duration of 15 s, and vacuum pressure of ±150 mmHg
  Interventions: Device: Conventional tracheal suctioning
- mechanical insufflation exsufflation (Experimental): The mechanical insufflation-exsufflation will be performed with the which will be applied 5 times in 5cough cycles in automatic mode, with insufflation and exsufflation pressures of + 40/-40 cmH2O, respectively. The duration of each phase was 3 s, without pause, and tracheal suctioning will be performed at the end of the procedure. Hyperoxygenation (100% O2) will be performed for 1 min before applying each technique and a 20 s interval will be allowed between repetitions. The secretion collected after each procedure will be stored in a disposable bronchial secretion collector for later weighing
  Interventions: Device: Mechanical insufflation/exsufflation

INTERVENTIONS:
Device: Conventional tracheal suctioning — Group 1 allocated to conventional tracheal suctioning,all patiemts will be followed up until discharge from ICU or death
  Tracheal suctioning will be performed following the American Association for Respiratory Care recommendations.
  Arms: Conventional endotracheal suctioning
Device: Mechanical insufflation/exsufflation — Group 2 will be allocated to mechanical insufflation-exsufflation which will be performed with the which will be applied 5 times in 5cough cycles in automatic mode, with insufflation and exsufflation pressures of + 40/-40 cmH2O, respectively. The duration of each phase was 3 s, without pause. Hyperoxygenation (100% O2) will be performed for 1 min before applying each technique and a 20 s interval will be allowed between repetitions.
  Arms: mechanical insufflation exsufflation

SUMMARY:
Aspiration of respiratory secretions is a frequently needed procedure in intubated patients .

Cough is an important defence mechanism to clear mucus from the upper and lower airways . The presence of an endotracheal tube impairs the ability to cough.There are a number of techniques to mobilise sputum and optimise airway clearance for invasively ventilated patients. Endotracheal suctioning is the most common intervention used to remove retained airway secretions from within the endotracheal tube, trachea and upper airways .Mechanical insufflation-exsufflation (MI-E) aids sputum clearance from upper and lower airways. This technique augments inspiratory and expiratory flows to improve sputum mobilisation, through the application of rapidly alternating positive and negative pressure, which approximates a normal cough

DETAILED DESCRIPTION:
Critically ill patients under invasive ventilation are at risk for sputum retention . Aspiration of respiratory secretions is a frequently needed procedure in intubated patients .

Cough is an important defence mechanism to clear mucus from the upper and lower airways . The presence of an endotracheal tube impairs the ability to cough. This prevents the enhancement of cough velocity . Furthermore, critically ill patients frequently have an impaired or no cough reflex due to depressed levels of consciousness, sedation, muscle weakness or muscle paralysis. Sputum retention, resulting from an inability to cough effectively, is one cause of extubation failure which in turn is associated with increased mortality.

There are a number of techniques to mobilise sputum and optimise airway clearance for invasively ventilated patients. Endotracheal suctioning is the most common intervention used to remove retained airway secretions from within the endotracheal tube, trachea and upper airways . Endotracheal suctioning though is not effective for clearing secretions from the lower airways .

New technologies and advanced methods have been developed to increase the effectiveness of mucus clearance in patients with acute respiratory failure, including mechanical insufflation-exsufflation devices. This technique has been described as an effective aid for mucus clearance in patients with chronic muscle weakness or neuromuscular disease.

Mechanical insufflation-exsufflation (MI-E) aids sputum clearance from upper and lower airways. This technique augments inspiratory and expiratory flows to improve sputum mobilisation, through the application of rapidly alternating positive and negative pressure, which approximates a normal cough .

ELIGIBILITY:
Inclusion Criteria:

Adult patients of both sexes on mechanical ventilation in RICU with any respiratory disease

Mechanically ventilated Patients without facial trauma

Mechanically ventilated Patients hemodynamically stable

Exclusion Criteria:

Patients diagnosed with barotrauma

Patients diagnosed with pneumothorax

History of bullous emphysema Known susceptibility to pneumothorax or pneumo-mediastinum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Assess effects of MIE on Volume of Secretions | 1 year
  Volume of Secretions measured in ml
Assess effects of MIE on respiratory rate | 1 year
  Respiratory rate measured by breaths per minute
Assess effects of MIE on tidal volume | 1 year
  Tidal volume measured in cubic centimeter
Assess effects of MIE on minute ventilation | 1 year
Assess effects of MIE on Oxygen saturation | 1 year
Assess effects of MIE on heart rate | 1 year
  Heart rate measured by beats per minute
Assess effects of MIE on blood pressur | 1 year
  Blood pressure measuered in mmHg

SECONDARY OUTCOMES:
Assess safety of Mechanical insufflation-exsufflation | 1 year
  assess safety according to number of complications e.g (hypotension, arrythmias, oxygen desaturaion, pneumothorax) and number of participants with complications

OTHER OUTCOMES:
Compare the effects and safety of MIE versus Endotracheal Suctioning | 1 year
  Comparison accoring to number of complications with each procedure

CONTACTS AND LOCATIONS:
Overall Officials: Reham Mohammed Elmorshedy, Principal Investigator — Assiut University; Marawan NaerELdin Mohammed, Principal Investigator — Assiut University

REFERENCES:
- [Background] Fahy JV, Dickey BF. Airway mucus function and dysfunction. N Engl J Med. 2010 Dec 2;363(23):2233-47. doi: 10.1056/NEJMra0910061. No abstract available. PMID 21121836
- [Background] American Association for Respiratory Care. AARC Clinical Practice Guidelines. Endotracheal suctioning of mechanically ventilated patients with artificial airways 2010. Respir Care. 2010 Jun;55(6):758-64. PMID 20507660
- [Background] McCool FD. Global physiology and pathophysiology of cough: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):48S-53S. doi: 10.1378/chest.129.1_suppl.48S. PMID 16428691
- [Background] Rothaar RC, Epstein SK. Extubation failure: magnitude of the problem, impact on outcomes, and prevention. Curr Opin Crit Care. 2003 Feb;9(1):59-66. doi: 10.1097/00075198-200302000-00011. PMID 12548031
- [Background] Sole ML, Bennett M, Ashworth S. Clinical Indicators for Endotracheal Suctioning in Adult Patients Receiving Mechanical Ventilation. Am J Crit Care. 2015 Jul;24(4):318-24; quiz 325. doi: 10.4037/ajcc2015794. PMID 26134331
- [Background] Ferreira de Camillis ML, Savi A, Goulart Rosa R, Figueiredo M, Wickert R, Borges LGA, Galant L, Teixeira C. Effects of Mechanical Insufflation-Exsufflation on Airway Mucus Clearance Among Mechanically Ventilated ICU Subjects. Respir Care. 2018 Dec;63(12):1471-1477. doi: 10.4187/respcare.06253. Epub 2018 Jul 17. PMID 30018175
- [Background] Chatwin M, Ross E, Hart N, Nickol AH, Polkey MI, Simonds AK. Cough augmentation with mechanical insufflation/exsufflation in patients with neuromuscular weakness. Eur Respir J. 2003 Mar;21(3):502-8. doi: 10.1183/09031936.03.00048102. PMID 12662009
- [Background] Vianello A, Corrado A, Arcaro G, Gallan F, Ori C, Minuzzo M, Bevilacqua M. Mechanical insufflation-exsufflation improves outcomes for neuromuscular disease patients with respiratory tract infections. Am J Phys Med Rehabil. 2005 Feb;84(2):83-8; discussion 89-91. doi: 10.1097/01.phm.0000151941.97266.96. PMID 15668554
- [Background] Chatwin M, Toussaint M, Goncalves MR, Sheers N, Mellies U, Gonzales-Bermejo J, Sancho J, Fauroux B, Andersen T, Hov B, Nygren-Bonnier M, Lacombe M, Pernet K, Kampelmacher M, Devaux C, Kinnett K, Sheehan D, Rao F, Villanova M, Berlowitz D, Morrow BM. Airway clearance techniques in neuromuscular disorders: A state of the art review. Respir Med. 2018 Mar;136:98-110. doi: 10.1016/j.rmed.2018.01.012. Epub 2018 Feb 6. PMID 29501255